CLINICAL TRIAL: NCT07062601
Title: Effect of Etomidate and Esketamine on Postoperative Pain After Tonsillectomy Undergoing Children With General Anesthesia
Brief Title: Etomidate and Esketamine on Postoperative Pain After Tonsillectomy Undergoing Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Xuzhang0109
Record Dates: First submitted 2025-06-29; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Etomidate; Esketamine; Tonsillectomy; Children
Keywords: Etomidate; Esketomine; Tonsillectomy
MeSH Terms: interventions — Etomidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etomidate and fentanyl group (Experimental): In the etomidate-fentanyl group (group A), 0.3 mg/kg etomidate and 4 µg/kg fentanyl were given at the induction of anesthesia, followed by continuous infusion of propofol at 4-12 mg/kg/h and remifentanil at 3-6 µg/kg/h until the end of the surgery, respectively
  Interventions: Drug: Etomidate and fentanyl group
- Etomidate and esketamine group (Experimental): In the etomidate-esketamine group (group B), induction of anesthesia with 0.3 mg/kg etomidate and 0.5 mg/kg esketamine , followed by continuous infusion of propofol at 4-12 mg/kg/h and remifentanil at 3-6 µg/kg/h until the end of the operation
  Interventions: Drug: Etomidate and esketamine group

INTERVENTIONS:
Drug: Etomidate and fentanyl group — In the etomidate-fentanyl group (group A), 0.3 mg/kg etomidate and 4 µg/kg fentanyl were given at the induction of anesthesia, followed by continuous infusion of propofol at 4-12 mg/kg/h and remifentanil at 3-6 µg/kg/h until the end of the surgery, respectively.
  Arms: Etomidate and fentanyl group
Drug: Etomidate and esketamine group — In the etomidate-esketamine group (group B), induction of anesthesia with 0.3 mg/kg etomidate and 0.5 mg/kg esketamine , followed by continuous infusion of propofol at 4-12 mg/kg/h and remifentanil at 3-6 µg/kg/h until the end of the operation
  Arms: Etomidate and esketamine group

SUMMARY:
Objective: To explore the effect of etomidate and esketamine on postoperative pain after tonsillectomy in children.

Methods: Investigators enrolled 64 children with American Society of Anesthesiologists (ASA) physical status I and II, aged 2-10 years, and scheduled for elective undergoing tonsillectomy with general anesthesia. All the enrolled patients were randomly divided into etomidate and fentanyl group (Group A) and etomidate and esketamine group (Group B). In the etomidate-fentanyl group (group A), 0.3 mg/kg etomidate and 4 µg/kg fentanyl were given at the induction of anesthesia, followed by continuous infusion of propofol at 4-12 mg/kg/h and remifentanil at 3-6 µg/kg/h until the end of the surgery, respectively; in the etomidate-esketamine group (group B), induction of anesthesia with 0.3 mg/kg etomidate and 0.5 mg/kg esketamine , followed by continuous infusion of propofol at 4-12 mg/kg/h and remifentanil at 3-6 µg/kg/h until the end of the operation. Anesthesiologists who were unaware of the grouping recorded the FlACC Pain Scale at 2 h, 8 h, and 24 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children who underwent elective tonsillectomy
* Aged 2-10 years old
* ASA class I-II

Exclusion Criteria:

* Children with hepatic or renal dysfunction
* Those with increased intracranial or intra-ocular pressure
* Children with schizophrenia, bipolar disorder, and any other psychiatric condition
* Children with preexisting chronic pain
* Children with preoperative combined sinus bradycardia or atrioventricular block

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
The face, legs, arms, crying, consolability (FLACC) pain scale | at 2 hours, 8 hours, and 24 hours after surgery
  Anesthesiologists who were unaware of the grouping recorded the face, legs, arms, crying, consolability (FLACC) pain scale at 2 hours, 8 hours, and 24 hours after surgery